CLINICAL TRIAL: NCT01423279
Title: The Effect of a Diabetic- and a Kidney-like Environment on Gene and Protein Expression in Mono- and Co-cultured Endothelial and Smooth Muscle Cells
Brief Title: The Effect of a Diabetic- and a Kidney-like Environment on Gene and Protein Expression in Cultured EC and SMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC11-0074CTIL; 0074-11-MMC (Other: Meir Medical Center , Israel)
Record Dates: First submitted 2011-08-24; First posted 2011-08-25 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Endothelial Dysfunction; Disorder of Smooth Muscle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This research is NOT part of an interventional trial, however the investigators use umbilical cord after birth for isolating endothelial and smooth muscle cells for academic research.

DETAILED DESCRIPTION:
Isolation and culturing of endothelial and smooth muscle muscles for academic research

ELIGIBILITY:
Inclusion Criteria:

* normal pregnancy

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women after normal birth
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The effect of a Diabetic- and a Kidney-like environment on gene and protein expression in mono- and co-cultured endothelial and smooth muscle cells | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Benchetrit, MD, Study Director — Nephrology dept. Meir Medical Center, Kfar Saba , Israel
Locations (1):
- Laboratory of Renal Physiology, Meir Medical Center ,, Kfar Saba, Israel

REFERENCES:
- [Background] Zitman-Gal T, Green J, Pasmanik-Chor M, Oron-Karni V, Bernheim J. Endothelial pro-atherosclerotic response to extracellular diabetic-like environment: possible role of thioredoxin-interacting protein. Nephrol Dial Transplant. 2010 Jul;25(7):2141-9. doi: 10.1093/ndt/gfp768. Epub 2010 Jan 19. PMID 20089511
- [Background] Talmor-Barkan Y, Bernheim J, Green J, Benchetrit S, Rashid G. Calcitriol counteracts endothelial cell pro-inflammatory processes in a chronic kidney disease-like environment. J Steroid Biochem Mol Biol. 2011 Mar;124(1-2):19-24. doi: 10.1016/j.jsbmb.2011.01.001. Epub 2011 Jan 12. PMID 21236342
- [Background] Talmor-Barkan Y, Rashid G, Weintal I, Green J, Bernheim J, Benchetrit S. Low extracellular Ca2+: a mediator of endothelial inflammation. Nephrol Dial Transplant. 2009 Nov;24(11):3306-12. doi: 10.1093/ndt/gfp354. Epub 2009 Jul 18. PMID 19617602
- [Background] Rashid G, Plotkin E, Klein O, Green J, Bernheim J, Benchetrit S. Parathyroid hormone decreases endothelial osteoprotegerin secretion: role of protein kinase A and C. Am J Physiol Renal Physiol. 2009 Jan;296(1):F60-6. doi: 10.1152/ajprenal.00622.2007. Epub 2008 Oct 22. PMID 18945829